CLINICAL TRIAL: NCT01957735
Title: A Phase 1a/b Non-randomized, Dose Escalation Study of the Safety, Pharmacokinetics, and Pharmacodynamics of Sterile BPM31510 (Ubidecarenone, USP) Nanosuspension Injection Administered Intravenously to Patients With Solid Tumors
Brief Title: BP31510 (Ubidecarenone,USP) Nanosuspension for Intravenous Injection to Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BPGbio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BP-31510IV-04
Record Dates: First submitted 2013-08-09; First posted 2013-10-08 (Estimated); Last update posted 2025-02-19 (Actual); Status verified 2019-11

CONDITIONS: Metastatic Cancer; Cancer; Solid Tumor
Keywords: metastatic cancer; solid tumor; unresectable tumor; brain cancer; lymphoma
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms; Brain Neoplasms; Lymphoma | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- BP31510 monotherapy (Experimental): * Starting dose level of BPM31510 will be 66 mg/kg administered by IV infusion over 48 hours 2 times per week of each 28-day cycle.The 2 doses will be administered over 4 consecutive days.The study drug will be administered undiluted via a central venous access device and the infusion rate will be controlled by a programmable ambulatory infusion pump.
  * first dose of each week of the cycle a loading dose will be infused over 1 hour with the remainder of the dose volume infused over 47 hours.At each dose level of Arm 1 and Arm 2, patients will be treated for either 8 hours at minimum of outpatient monitoring or inpatient monitoring for the first 24-hrs of the first infusion of Cycle 1.
  * second dose of each week of the cycle, the total dose volume given over 48 hours with no loading dose.
  Interventions: Drug: BP31510 monotherapy
- BP31510 in combination with chemotherapy (Active Comparator): standard 3+3 design will be used for Arm 2 of the study. BPM31510 will be started at one dose level below the dose that has been studied and determined to be safe in the monotherapy portion of the trial. Arm 2 patients will be enrolled onto one of 3 chemotherapies, gemcitabine, 5-FU, or docetaxel according to the dose levels below:
  * Gemcitabine IV once weekly at a starting dose of 600 mg/m2 ;
  * 5-Fluorouracil (5-FU) IV once weekly at a starting dose of 350 mg/m2 with leucovorin (LV) 100 mg/m2; OR
  * Docetaxel IV once weekly at a starting dose of 20 mg/m2.
  * Note:Both BPM31510 and the chemotherapy agent can escalate simultaneously in Cohorts 3 and 4 only if there are no DLTs observed in the previous cohorts. If one or more DLTs are observed, then intermediate dose levels will be added where one agent is escalated.
  Interventions: Drug: BP31510 in combination with chemotherapy

INTERVENTIONS:
Drug: BP31510 monotherapy
  Arms: BP31510 monotherapy
Drug: BP31510 in combination with chemotherapy
  Arms: BP31510 in combination with chemotherapy

SUMMARY:
This is a Phase 1a/b multicenter, open-label, non-randomized, dose-escalation study to examine the dose limiting toxicities (DLT) of BPM31510 administered as a 144-hour continuous intravenous (IV) infusion as monotherapy(treatment Arm 1) and in combination with chemotherapy (treatment Arm 2) in patients with solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1a/b multicenter, open-label, non-randomized, dose-escalation study to examine the dose limiting toxicities (DLT) of BPM31510 administered as a 144-hour continuous intravenous (IV) infusion as monotherapy(treatment Arm 1)and in combination with chemotherapy (treatment Arm 2) in patients with solid tumors.In the Phase 1a portion of the trial, patients who meet eligibility parameters will receive 2 consecutive 72-hour infusions of BPM31510 twice weekly on Tuesday and Friday (i.e., Days 1, 4, 8, 11, 18, 22 and 25), essentially receiving BPM31510 treatment for 144 hours per week of each 28-day cycle. At each dose level of Arm 1 and Arm 2, patients will be treated for either 8 hours at minimum of outpatient monitoring or inpatient monitoring for the first 24-hrs of the first infusion of Cycle 1.All other treatments will be administered in an outpatient setting.Dose limiting toxicities will be assessed during Cycle 1.

The study is a standard 3 + 3 dose escalation design with the dose escalated in successive cohorts of 3 to 6 patients each.Toxicity at each dose level will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE v4.02). Safety oversight will be provided by the Cohort Review Committee (CRC).The CRC will review and confirm all DLTs and will continue to monitor safety throughout the study (including Arm 2).

Assessments of the antitumor activity of BPM31510 will be performed at the end of Cycle 2 and every 2 cycles thereafter using standard techniques such as computerized tomography (CT) or magnetic resonance imaging (MRI) for patients with measurable disease.Response will be evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 .Patients who experience no unacceptable toxicity or disease progression, may receive additional 28-day cycles for up to 1 year on Arm 1 or 2. Patients on Arm 1 who progress may elect to continue BPM31510 treatment in combination with gemcitabine, 5-FU, or docetaxel at the treating physician's discretion. Once a dose level of BPM31510 monotherapy is evaluated and the CRC determines it safe to escalate to the next dose level, Cohort 1 of Treatment Arm 2 of BPM31510 in combination with chemotherapy will open to accrual. Cohort 1 of Arm 2 patients will be enrolled onto one of 3 chemotherapies, gemcitabine, 5-FU, or docetaxel. Cycle 1 of combination therapy (Arm 2) is 6 weeks in duration for patients with BPM31510 administered twice weekly on Tuesday and Friday for 6 weeks and chemotherapy administered on Mondays, Days 21, 28 and 35. Cycles 2-12 are 4 weeks in duration with BPM31510 administered twice weekly on Tuesday and Friday for 4 weeks and chemotherapy administered on Mondays, Days 7, 14 and 21. Dose limiting toxicities will be assessed during Cycle 1. Response will be assessed after Cycle 2 (10 weeks) and responders who continue onto Cycles 2-12 will be assessed every 2 cycles (8 weeks). Patients who progress and crossover to Arm 2 will be reconsented and must meet eligibility before restarting BPM31510. Crossover patients are not evaluated for DLTs on Arm 2 and all cycles of combination therapy are 4 weeks in duration (Cycles 1-12). BPM31510 is administered twice weekly on Tuesdays and Fridays for 4 weeks and chemotherapy administered on Mondays, Days 7, 14 and 21 for all crossover patients on Arm 2. Patients will continue BPM31510 in combination with chemotherapy for a maximum of 12 cycles in the absence of intolerable toxicity and progression. Patients on Arm 2 who progress on one type of chemotherapy may not switch to one of the other chemotherapy agents in combination with BPM31510.However, if the chemotherapy component (ie, 5-FU, gemcitabine, or docetaxel) of combination therapy is discontinued due to chemotherapy-related toxicity, patients may continue to receive BPM31510 as monotherapy.

Once the maximum tolerated dose (MTD) of BPM31510 as monotherapy and in combination with chemotherapy are established, an expansion cohort will be enrolled (a total of 12-15 patients for monotherapy and a total of 10 patients for each combination therapy).

ELIGIBILITY:
Inclusion Criteria:

* The patient has a histologically confirmed solid tumor that is metastatic or unresectable for which standard measures do not exist or are no longer effective. (Patients with primary brain cancer or lymphoma are permitted. Patients with brain metastases are allowed if whole brain radiation was performed and is documented stable for ≥ 6 weeks)
* The patient is at least 18 years old.
* The patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* The patient has a life expectancy of > 3 months.
* Sexually active patients and their partners agree to use an accepted method of contraception during the course of the study
* Female patients of childbearing potential must have a negative pregnancy test within 1 week prior to beginning study treatment.
* The patient has adequate organ and marrow function as follows:
* ANC ≥ 1500 mm3, platelets ≥ 100,000/mm3, hemoglobin ≥ 9 g/dL,
* serum creatinine ≤1.8 mg/dL or creatinine clearance > 50 mL/min (Appendix I);
* bilirubin ≤ 1.5 mg/dL; alanine aminotransferase (ALT), aspartate transaminase (AST) ≤ 2.5 times the upper limit of normal if no liver involvement or ≤ 5 times the upper limit of normal with liver involvement.
* The patient has serum electrolytes (including calcium, magnesium, phosphorous, sodium and potassium) within normal limits (supplementation to maintain normal electrolytes is allowed).
* The patient has adequate coagulation: prothrombin time (PT), partial thromboplastin time (PTT), and an International Normalized Ratio within normal limits.
* The patient is capable of understanding and complying with the protocol and has signed the informed consent document.

Exclusion Criteria:

* The patient has uncontrolled intercurrent illness including, but not limited to uncontrolled infection, symptomatic congestive heart failure (NYHA class III and IV), uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* The patient has active heart disease including myocardial infarction within previous 3 months, symptomatic coronary artery disease, arrhythmias not controlled by medication, unstable angina pectoris, or uncontrolled congestive heart failure (NYHA class III and IV)
* The patient has received chemotherapy or radiotherapy within 4 weeks or has received nitrosoureas or mitomycin C within 6 weeks prior to the first dose of study drug.
* The patient has received radiation to ≥ 25% of his or her bone marrow within 4 weeks of the first dose of study drug.
* The patient has received an investigational drug within 30 days of the first dose of study drug.
* The patient has not recovered to grade ≤ 1 adverse events (AEs) due to investigational drugs or other medications, administered more than 2 weeks prior to the first dose of study drug, with the exception of neurotoxicity attributed to oxaliplatin or taxanes, which must have recovered to < 2 prior to study initiation.
* The patient is pregnant or lactating.
* The patient is known to be positive for the human immunodeficiency virus (HIV). The effect of BPM31510 on HIV medications is unknown. Note: HIV testing is not required for eligibility, but if performed previously and was positive, the patient is ineligible for the study.
* The patient has an inability or unwillingness to abide by the study protocol or cooperate fully with the investigator or designee.
* The patient is receiving digoxin, digitoxin, lanatoside C or any type of digitalis alkaloids.
* The patient is receiving colony stimulating factors (CSFs) that cannot be held during the monitoring period for dose-limiting toxicities (DLT).
* The patient has uncontrolled or severe coagulopathies or a history of clinically significant bleeding within the past 6 months, such as hemoptysis, epistaxis, hematochezia, hematuria, or gastrointestinal bleeding.
* The patient has a known predisposition for bleeding such as von Willebrand's disease or other such condition.
* The patient requires therapeutic doses of any anticoagulant, including LMWH. Concomitant use of warfarin, even at prophylactic doses, is prohibited.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2013-10; Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Determine Maximum Tolerated Dose (MTD) of BP31510 | Wach week of treatment for the duration of Cycle 1 up to 4 weeks on Arm 1 and 6 weeks for Arm 2
  Dose limiting toxicities will be assessed during Cycle 1 (first four weeks of Arm 1 and 6 weeks for Arm 2) of the study. Blood samples for pharmacokinetic and pharmacodynamic analyses will be collected during each cycle of monotherapy and combination therapy. Urine samples for determination of BPM31510 renal clearance will be collected only during Cycle 1 of monotherapy and combination therapy. A PET scan will be performed within 2 weeks prior to starting treatment and after 2 weeks of BPM31510 treatment, and 8 weeks of treatment on Arm 1 or 10 weeks of treatment on Arm 2. Core biopsies (2-3) will be performed at the time of baseline and Week 2 PET scan for patients who opt-in to participate in these exploratory studies.

SECONDARY OUTCOMES:
To evaluate plasma pharmacokinetics (PK) of BPM31510 | Each cycle (every 4 weeks) for for up to 1 year
  To evaluate plasma pharmacokinetics (PK) of BPM31510 monotherapy and BPM31510 in combination with chemotherapy when administered as a 144-hour IV infusion in patients with solid tumors.
  Blood samples for pharmacokinetic and pharmacodynamic analyses will be collected during each cycle of monotherapy and combination therapy. Urine samples for determination of BPM31510 renal clearance will be collected only during Cycle 1 of monotherapy and combination therapy. A PET scan will be performed within 2 weeks prior to starting treatment and after 2 weeks of BPM31510 treatment, and 8 weeks of treatment on Arm 1 or 10 weeks of treatment on Arm 2. Core biopsies (2-3) will be performed at the time of baseline and Week 2 PET scan for patients who opt-in to participate in these exploratory studies.
To estimate renal clearance of BPM31510 | Each cycle (every 4 weeks) for for up to 1 year
  To estimate renal clearance of BPM31510 monotherapy and BPM31510 in combination with chemotherapy when administered as a 144-hour IV infusion in patients with solid tumors
  Blood samples for pharmacokinetic and pharmacodynamic analyses will be collected during each cycle of monotherapy and combination therapy. Urine samples for determination of BPM31510 renal clearance will be collected only during Cycle 1 of monotherapy and combination therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Manish A Shah, MD, Principal Investigator — Weill Cornell Solid Tumor Oncology Practice; Vivek Subbiah, MD, Principal Investigator — M.D. Anderson Cancer Center; Kim-Son Nguyen, MD, Principal Investigator — Palo Alto Medical Foundation
Locations (3):
- United States (3):
  - Palo Alto Medical Foundation, Sunnyvale, California
  - Weill Cornell Solid Tumor Oncology Practice, New York, New York
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No